CLINICAL TRIAL: NCT03486730
Title: A Cancer Research UK Phase I/IIa Clinical Trial of BT1718, (A Bicycle Drug Conjugate) Given Intravenously in Patients with Advanced Solid Tumours.
Brief Title: BT1718 in Patients with Advanced Solid Tumours.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: Bicycle Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/17/009; 2016-004633-24 (EudraCT Number)
Record Dates: First submitted 2018-01-18; First posted 2018-04-03 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumours; Non-Small Cell Lung Cancer; Non-Small Cell Lung Sarcoma; Oesophageal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose escalation phase (Experimental): Groups of patients will receive increasing doses of BT1718 to find a safe dose that best targets the cancer cells. In this phase it is expected that approximately 50-60 patients with advanced solid tumours will be entered in the study.
  Interventions: Drug: BT1718
- Dose expansion phase (Experimental): Larger groups of patients will receive the selected dose of BT1718 to allow us to find out more about how the drug is working. In this phase it is proposed that up to 70 patients with tumour types known to commonly overexpress MT1-MMP and where MT1-MMP overexpression is confirmed during prospective and retrospective (in appropriate patients) selection at enrolment (i.e. squamous non-small cell lung cancer) will be entered in the study.
  Interventions: Drug: BT1718

INTERVENTIONS:
Drug: BT1718 — Dose escalation will consist of Stage 1 and 2. Stage 1 patients will receive BT1718 intravenously twice a week (D: 1,4,8,11,15,18) for 3 out of 4 weeks. Starting dose will be 0.6mg/m2. Single patient cohorts will be explored, but it will change to 3 to 6 patients cohorts. Stage 2 patients will receive BT1718 intravenously once a week (D: 1,8,15) for 3 out of 4 weeks. This stage will have 3 to 6 patient cohorts until the recommended dose is established. The expansion phase will consist of two or more expansion cohorts to include tumour types known to commonly over-express MT1-MMP and where MT1-MMP overexpression is confirmed during prospective and retrospective (in appropriate patients) selection at enrolment. A squamous NSCLC and basket cohort will include approximately 16 patients each with high MT1-MMP levels. In the expansion cohorts BT1718 will be administered intravenously at the once weekly RP2D established in Phase I, Stage 2.

SUMMARY:
This clinical trial is looking at a drug called BT1718 in adult patients with advanced solid tumours. The main aim of the study is to find the maximum dose of BT1718 that can be given safely to patients; learn more about the potential side effects of BT1718 and how they can be treated and also what happens to BT1718 inside the body.

DETAILED DESCRIPTION:
BT1718 is a type of drug called a 'bicycle drug conjugate' which is designed to target and inhibit the function of the protein 'membrane type 1 metalloproteinase' (MT1-MMP). MT1-MMP is involved in breaking down the proteins that usually surround a cell; however in cancer cells it can allow a cancer to grow and spread. MT1-MMP is usually found at a low level in normal cells, but can reach higher levels in cancer cells.

BT1718 has been designed to recognise and attach itself to the MT1-MMP protein. Once attached a segment of BT1718 is taken into the cancer cell which causes it to die (DM1 toxin).

This is a first in human clinical study which has two phases. A 'dose escalation' phase where groups of patients will receive increasing doses of BT1718 to find a safe dose that best targets the cancer cells. In this phase it is expected that approximately 50-60 patients with advanced solid tumours will be entered in the study.

An 'expansion phase' where larger groups of patients will receive the selected dose of BT1718 to allow us to find out more about how the drug is working. In this phase at the optimal dose/schedule(s), patients will be enrolled with tumour types known to commonly overexpress MT1-MMP and where MT1-MMP overexpression is confirmed during prospective and retrospective (in appropriate patients) selection at enrolment (i.e. squamous non-small cell lung cancer). It is expected that up to an additional 70 patients will be required to complete this phase.

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up
2. Phase I, dose escalation phase (Stages 1 and 2):

   • Histologically or cytologically proven advanced solid tumour, refractory to conventional treatment, or for which no conventional therapy is considered appropriate by the Investigator or is declined by the patient.

   Phase IIa, expansion phase:
   * Histologically or cytologically proven advanced solid tumour of particular interest based on pre-clinical and clinical data, refractory to conventional treatment, or for which no conventional therapy is considered appropriate by the Investigator or is declined by the patient. Phase IIa expansion cohorts will be:

     1. Squamous NSCLC cohort - retrospective MT1-MMP testing.
     2. Basket cohort (advanced solid tumours, excluding patients eligible for one of the other recruiting expansion cohorts) - high MT1-MMP expression by IHC assay using archival tumour sample (mandatory fresh tumour samples for those patients without available archival tumour samples or additional analysis is deemed necessary). Retrospective testing may be permitted for tumour types estimated to have high MT1-MMP positivity rates as per the Laboratory manual.
     3. Additional expansion cohort(s) of squamous oesophageal cancer if confirmed as recruiting by the Sponsor.
   * At least one measurable lesion according to RECIST criteria Version 1.1, that has had objective radiological progression on or after the last therapy.
   * Consent for pre-treatment and post-treatment fresh tumour biopsy sample in a minimum of eight patients in the squamous NSCLC cohort, squamous oesophageal cohort (if confirmed as recruiting by the Sponsor) and all patients in the basket cohort (except patients with a very high MT1-MMP H-score if agreed with the Sponsor and PI as defined in the Laboratory Manual).
   * Consent for pre-treatment and post-treatment non-tumour sample (optional) for patients having a pre and post treatment tumour biopsy.
   * Consent for pre and post treatment skin punch biopsy (optional).
3. Life expectancy of at least 12 weeks.
4. World Health Organisation (WHO) performance status of 0 - 1.
5. Haematological and biochemical indices within the ranges shown below. These measurements should be performed to confirm the patient's eligibility.

   Haemoglobin (Hb): ≥90.0 g/L, or ≥100.0 g/L if transfusion within last four weeks Absolute neutrophil count (ANC): ≥1.5 x 10^9/L Platelet count: ≥100 x 10^9/L Bilirubin: ≤1.5 x upper limit of normal (ULN). NB: >1.5 ULN, acceptable if conjugated bilirubin is ≤1.5x ULN Alanine amino-transferase (ALT), aspartate amino-transferase (AST) and alkaline phosphatase (ALP) and gamma-glutamyl transferase (GGT) : ≤2.5 x ULN (or ≤5 x ULN if has liver metastases) Renal function

   Either:

   Serum creatinine: ≤1.5 x ULN

   Or:

   Calculated creatinine clearance (using the Wright or Cockcroft & Gault [C&G] formula): GFR ≥50 mL/min (uncorrected value)

   Or:

   Isotope clearance measurement: GFR ≥50 mL/min (corrected value)
6. 16 years or over at the time consent is given
7. Consent to access and analyse any available archival tissue.

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), systemic anti-cancer therapy (with the exception of life-long hormone suppression such as LHRH agents in prostate cancer) or investigational medicinal products during the previous four weeks (six weeks for nitrosoureas, mitomycin-C) before treatment (or first dose of an immunotherapy during the previous 12 weeks).
2. Prior bone marrow transplant, myeloablative conditioning, or extensive radiotherapy to greater than 25% of bone marrow, within previous eight weeks of first BT1718 dose.
3. Ongoing toxic manifestations of previous treatments greater than NCI CTCAE Grade 1. Exceptions to this are alopecia, amenorrhea/oligospermia and any other ongoing toxic manifestation which in the opinion of the Investigator and the Medical Advisor should not exclude the patient.
4. Any CNS metastases (unless had local therapy and are asymptomatic and radiologically-stable off steroids for the last four weeks).
5. Current or prior malignancy which could affect compliance with the protocol or interpretation of results. Patients with curatively-treated non-melanoma skin cancer, non-muscle-invasive bladder cancer, or carcinomas-in-situ are generally eligible.
6. Female patients who are able to become pregnant (or are already pregnant or lactating). However, those patients who have a negative serum or urine pregnancy test before enrolment and agree to use two forms of contraception (one effective form plus a barrier method) [oral, injected or implanted hormonal contraception and condom; intra-uterine device and condom; diaphragm with spermicidal gel and condom] or agree to sexual abstinence, effective from the first administration of BT1718, throughout the trial and for six months afterwards are considered eligible.
7. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using a barrier method of contraception [condom plus spermicide] or to sexual abstinence effective from the first administration of BT1718, throughout the trial and for six months afterwards. Men with partners of child-bearing potential must also be willing to ensure that their partner uses an effective method of contraception for the same duration for example, hormonal contraception, intrauterine device, diaphragm with spermicidal gel or sexual abstinence). Men with pregnant or lactating partners must be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure of the foetus or neonate.
8. Surgery from which the patient has not yet recovered.
9. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
10. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
11. Patients with significant cardiovascular disease are excluded as defined by:

    1. Current congestive heart failure requiring therapy (NYHA III or IV - Appendix 3) or known LVEF <40% (moderate to severe)
    2. History of unstable angina pectoris or myocardial infarction up to six months prior to trial entry, or of current poorly controlled angina (symptoms weekly or more)
    3. Presence of symptomatic or severe valvular heart disease (severe by local echographic criteria or AHA/ACC Stage C or D - Appendix 4)
    4. History of a clinically significant cardiac arrhythmia up to six months prior to trial entry (asymptomatic atrial fibrillation or asymptomatic first-degree heart block are permitted)
12. Previous known allergy to one of the constituents or excipients of BT1718.
13. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I/IIa study of BT1718. Participation in an observational trial or interventional clinical trial which does not involve administration of an IMP and which would not place an unacceptable burden on the patient in the opinion of the Investigator and Medical Advisor would be acceptable.
14. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum dose | When sufficient patients have had the opportunity to complete 1 Cycle (28 days).
  Determine a dose at which no more than one out of six patients at the same dose level experiences a probable or highly probable BT1718-related dose limiting toxicity (DLT).
Determination of the frequency and causality of each adverse event | When sufficient patients have had the opportunity to complete 1 Cycle (28 days).
  Determine the frequency and causality of each adverse event (AE) to BT1718 and grade severity according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.02.

SECONDARY OUTCOMES:
Measurement of the maximum observed plasma concentration (Cmax) of BT1718 in plasma, both as an intact and cleaved molecule. | Up to 24 timepoints from the first dose of BT1718 over the first two cycles (i.e. Cycle 1 and Cycle 2). Each Cycle is 28 days.
  Measurement of the maximum observed plasma concentration (Cmax) of BT1718 in plasma, both as an intact and cleaved molecule.
Measurement of the area under the curve (AUC) of BT1718 in plasma, both as an intact and cleaved molecule. | Up to 24 timepoints from the first dose of BT1718 over the first two cycles (i.e. Cycle 1 and Cycle 2). Each Cycle is 28 days.
  Measurement of the area under the curve (AUC) of BT1718 in plasma, both as an intact and cleaved molecule.
Measurement of the terminal elimination half-life (t½) of BT1718 in plasma, both as an intact and cleaved molecule. | Up to 24 timepoints from the first dose of BT1718 over the first two cycles (i.e. Cycle 1 and Cycle 2). Each Cycle is 28 days.
  Measurement of the terminal elimination half-life (t½) of BT1718 in plasma, both as an intact and cleaved molecule.
Measurement of other PK parameters of BT1718 in plasma, both as an intact and cleaved molecule. | Up to 24 timepoints from the first dose of BT1718 over the first two cycles (i.e. Cycle 1 and Cycle 2). Each Cycle is 28 days.
  Measurement of other PK parameters of BT1718 in plasma, both as an intact and cleaved molecule.
Assess anti-tumour response according to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 using computerised tomography (CT) or magnetic resonance imaging (MRI) scans. | Evaluation will be at database lock - 4 weeks after the last patient last visit
  Assess anti-tumour response according to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 using computerised tomography (CT) or magnetic resonance imaging (MRI) scans.
Estimate progression-free survival | Evaluation will be at database lock - 4 weeks after the last patient last visit
  Estimate progression-free survival
Estimate progression-free survival rate at six months | Six months
  Estimate progression-free survival rate at six months
Estimate overall survival | Evaluation will be at database lock - 4 weeks after the last patient last visit
  Estimate overall survival
Estimate duration of response | Evaluation will be at database lock - 4 weeks after the last patient last visit
  Estimate duration of response

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrookes Hospital, Cambridge
  - The Beatson Hospital, Glasgow
  - Royal Marsden Hospital and The Institute of Cancer Research, London
  - University College London Hospital NHS Foundation Trust, London
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BT1718 ISRCTN Record (including basic results) — https://doi.org/10.1186/ISRCTN11160449